CLINICAL TRIAL: NCT00466791
Title: A Phase II, Randomized, Double-blind, Multi-center, Placebo-controlled, Dose Optimization, Analog Classroom, Crossover Study Designed to Assess the Time Course of Treatment Effect, Tolerability and Safety of Methylphenidate Transdermal System (MTS) in Pediatric Patients Aged 6-12 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Classroom Study to Assess Efficacy and Safety of MTS in Pediatric Patients Aged 6-12 With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD485-201
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate Transdermal System (Active Comparator): Transdermal patch, 27.5mg, 41.3mg, 55mg, and 82.5mg, daily for 11 weeks
  Interventions: Drug: Methylphenidate Transdermal System
- Placebo (Placebo Comparator): Transdermal patch, 0mg, daily for 11 weeks
  Interventions: Drug: Methylphenidate Transdermal System

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — Placebo
  Other Names: ADHD Patch

SUMMARY:
Evaluate the behavioral effects of MTS in children aged 6-12 with ADHD

DETAILED DESCRIPTION:
Evaluate the behavioral effects measured by the SKAMP deportment scale of MTS compared to placebo in children aged 6-12 with ADHD

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis ADHD
* Total score of greater than or equal to 26 on ADHD-RS-IV
* IQ of greater than or equal to 80
* Blood pressure measurements within 95th percentile for age, gender, height at screening and baseline

Exclusion Criteria:

* Current controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis (except ODD)
* Known nonresponder to psychostimulant treatment
* BMI for age greater than 90th percentile
* History of seizures during last 2 years
* Conduct Disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Score on SKAMP rating scale at 2,3,4.5,6,7.5,9,10.5 and 12 hours post application of MTS | 2,3,4.5,6,7.5,9,10.5 and 12 hours

SECONDARY OUTCOMES:
PERMP scores | pre-dose, 2.0, 3.0, 4.5, 6.0, 7.5, 9.0, 10.5 and 12.0 hours post application
Clinician-rated ADHD-RS-IV score | 2,3,4.5,6,7.5,9,10.5 and 12 hours
CGI-I score | Weeks 1-9
PGA | Weeks 1-9
CPRS-R score | Weeks 1-9

CONTACTS AND LOCATIONS:
Locations (1):
- UCI Child Development Center, Irvine, California, United States

REFERENCES:
- [Result] McGough JJ, Wigal SB, Abikoff H, Turnbow JM, Posner K, Moon E. A randomized, double-blind, placebo-controlled, laboratory classroom assessment of methylphenidate transdermal system in children with ADHD. J Atten Disord. 2006 Feb;9(3):476-85. doi: 10.1177/1087054705284089. PMID 16481664
- See also: FDA-approved labelling information, US only — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?CFID=20377655&CFTOKEN=caaa9085d296aa43-A8C6AE4E-1143-D1C5-FB7BD1C853149DF7
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html